CLINICAL TRIAL: NCT06822829
Title: Multicenter Retrospective Observational Study of Relapsed Diffuse Large B-Cell Lymphoma Presenting As Indolent Lymphoma
Acronym: REVERSE_2021
Status: Recruiting | Type: Observational
Sponsor: Azienda USL Reggio Emilia - IRCCS (Other Government)
Responsible Party: Sponsor
Other Study IDs: 446/2023/OSS/IRCCSRE
Record Dates: First submitted 2025-02-07; First posted 2025-02-12 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Diffuse Large B Cell Lymphoma (DLBCL); Indolent B-Cell Lymphomas; Indolent B Cell Lymphoma
Keywords: indolent relapse; diffuse large b cell lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients diagnosed with diffuse large B-cell lymphoma: Retrospective cohort of patients diagnosed with diffuse large B-cell lymphoma (DLBCL) who relapsed as indolent B-cell lymphoma between 2010 and 2020

SUMMARY:
Most relapses of diffuse large B-cell lymphoma (DLBCL) occur as high-grade lymphoma within the first two years after diagnosis. Relapses as indolent lymphoma are rare events, and the true incidence of this phenomenon is unknown, since literature data are scarce/ and usually restricted to case reports. Analogously, reported treatment strategies are rather heterogeneous, since no standard of care is established and advanced age together with previous anthracycline exposure may narrow the therapeutic choice.

The goal of this observational study is to assess epidemiological, clinical characteristics and survival of diffuse large b-cell lymphoma (DLBCL) relapsing as indolent lymphoma.

More precisely, the study aims at identifying diagnostic and imaging features associated with relapse as indolent lymphoma and at evaluating disease response to selected therapies.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older at the time of diagnosis.
* Previous diagnosis of diffuse large B-cell lymphoma with/without a discordant component of indolent B-cell lymphoma, or previous diagnosis of diffuse large B-cell lymphoma transformed from indolent B-cell lymphoma.
* First-line treatment for diffuse large B-cell lymphoma.
* Histologically documented relapse of indolent B-cell lymphoma, diagnosed between 2010 and 2020.
* Availability of the histological report of the relapse.
* Availability of clinical and laboratory data related to both the initial diagnosis and relapse.
* Availability of follow-up data.
* Consent to participate in the study and signing of the specific informed consent form (for living and/or contactable patients).

Exclusion Criteria:

- None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be proposed to patients diagnosed with diffuse large B-cell lymphoma (DLBCL) who have relapsed as indolent B-cell lymphoma, with a histologically confirmed diagnosis of relapse and availability of the histological report. Patients who are still alive will be contacted and informed by the specialist about the study's objectives and will be required to sign a specific informed consent form. For patients lost to follow-up or deceased, a waiver of informed consent has been obtained from the Ethics Committee in accordance with applicable regulations.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-08-19 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | Up to 2 years
  OS is calculated from the date of initiation of treatment for indolent lymphoma relapse to death from any cause or the last follow-up for censored cases.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | Up to 2 years
  PFS is measured from the date of initiation of treatment for indolent lymphoma relapse until disease progression or death, or the last follow-up for censored cases.
Response Rate | Up to 2 years
  Response to treatment for indolent B-cell lymphoma relapse will be assessed in terms of complete response, partial response, stable disease, and progression, according to the Lugano Classification criteria (Cheson B et al, JCO 2014).
Adverse Events | Up to 2 years
  Long-term adverse events occurring during follow-up (after treatment for indolent lymphoma relapse) will be categorized and graded according to the Common Toxicity Criteria for Adverse Events, referencing the most recent version available.
Type of Therapy | Up to 2 years
  Description of the therapeutic pathway adopted for first-line treatment of diffuse large B-cell lymphoma and second-line treatment for indolent lymphoma relapse.
Cause of Death | Up to 2 years
  Description of the causes of death, with particular focus on death due to disease progression versus other causes.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Elena Nizzoli, MD, Principal Investigator — Azienda USL - IRCCS di Reggio Emilia
Locations (1):
- Azienda USL IRCCS di Reggio Emilia, Reggio Emilia, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang Y, Link BK, Witzig TE, Maurer MJ, Allmer C, King RL, Feldman AL, Habermann TM, Ansell SM, Slager SL, Cerhan JR, Nowakowski GS. Impact of concurrent indolent lymphoma on the clinical outcome of newly diagnosed diffuse large B-cell lymphoma. Blood. 2019 Oct 17;134(16):1289-1297. doi: 10.1182/blood.2019000858. PMID 31350266
- [Background] Ghesquieres H, Berger F, Felman P, Callet-Bauchu E, Bryon PA, Traverse-Glehen A, Thieblemont C, Baseggio L, Michallet AS, Coiffier B, Salles G. Clinicopathologic characteristics and outcome of diffuse large B-cell lymphomas presenting with an associated low-grade component at diagnosis. J Clin Oncol. 2006 Nov 20;24(33):5234-41. doi: 10.1200/JCO.2006.07.5671. Epub 2006 Oct 16. PMID 17043351